CLINICAL TRIAL: NCT06461572
Title: Effects of Power Ball on Proximal Muscle Control and Refractive Error in Children With Developmental Delay
Brief Title: Effects of Power Ball on Proximal Muscle and Refractive Errors in Developmental Delay.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0790
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Developmental Delay
Keywords: Developmental delay; Refractive error; Power ball; Muscle control
MeSH Terms: conditions — Learning Disabilities; Refractive Errors | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. two groups of 7-12 years of age will be perform in which participants will be randomly divided. Group A will receive conventional therapy. Group B will receive Together with conventional treatment, this group will engage in power ball exercises for neck stability and strengthening.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (Active Comparator): This group will receive conventional therapy.
  Interventions: Other: conventional therapy
- conventional therapy with Standard therapy and stability exercises (Experimental): This group will receive conventional therapy with standard therapy and stability exercises.
  Interventions: Other: conventional therapy along with standard therapy and stability exercises.

INTERVENTIONS:
Other: conventional therapy — This group will receive conventional physiotherapy, which will consist of manual resistance-based neck strengthening exercises. The exercises will last 30 minutes apiece and cover cervical flexion, extension, side flexion, side flexion with rotation, and pure rotation with moderate resistance. The power ball's effect on proximal muscle control and refractive error in children with developmental delays will also be discussed.
  Arms: conventional therapy
Other: conventional therapy along with standard therapy and stability exercises. — Group B: In addition to standard care, this group will engage in power ball exercises for neck stability and strengthening. Gradually, the resistance will rise.
  Three mints in each position for a total of fifteen mints of ball exercises. At first, Powerball progressively strengthened the muscle and reduced the pain , and with continued development, allowed them to move in a pain-free range.
  Arms: conventional therapy with Standard therapy and stability exercises

SUMMARY:
When a child does not meet developmental milestones at the anticipated times, it is referred to as having a developmental delay. These benchmarks cover social, emotional, cognitive, physical, and communication abilities. Developmental delays can result from a number of factors, including genetic circumstances, early delivery, specific medical issues, or external variables. Although they mainly impair vision, refractive errors are unrelated to developmental delays. Because vision facilitates interaction with the environment, it is vital to a child's development. Early detection of uncorrected refractive defects and related vision loss in children can pose a challenge. To ascertain whether an increase is suitable and successful, a thorough evaluation of the child's readiness and the application of pertinent measurement techniques may be necessary. An analysis looks into Randomized Controlled Trial will be the type of study design used. There will be two groups of conveniently randomized sample size of thirty-two. The data analysis will be done using SPSS version 22.0. To verify normality, the Shapiro-Wilk test will be employed. The study will be carried out in the department of physical therapy of the rising sun and the Lahore rehab facility. The study will be finished six months from the time the synopsis is approved. A sample size of thirty-two was determined using the OPENEPI tool. The VQOL/item Tool and pediatric manual muscle testing will be used. For four weeks, the control group will receive standard physical therapy care. Group B: Experimental Group: For five weeks, a traditional physical therapy regimen and Powerball exercises will be administered.

DETAILED DESCRIPTION:
Group A: conventional physiotherapy will be administered to this group. Manual resistance exercises for neck strengthening are part of conventional physical therapy. Cervical flexion, extension, side flexion, side flexion with rotation, and pure rotation with mild resistance are the exercises used to strengthen the neck. There will be three 30-minute sessions. Strengthening will take place over the course of 15 mints.

Group B: In addition to standard care, this group will engage in power ball exercises for neck stability and strengthening. Gradually, the resistance will rise.

Three mints in each position for a total of fifteen mints of ball exercises. At first, Powerball reduced the pain, progressively strengthened them, and with continued development, allowed them to move in a pain-free range.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-12 years
* Both genders
* Children with refractive error
* Children with affected developmental delay

Exclusion Criteria:

* Any neurological condition (Epilepsy and seizures)
* Any congenital defects
* Genetic disorder
* Surgery in last 6 months

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
VQOL/ITEM Tool | 4 weeks
  The refractive errors and visual acuity of children who have developmental delays will be assessed using this tool. The ability of child to identify the size of the letters on a card held 20 feet (6 meters) away or on a standardized chart (Snellen chart). There will be specific charts used for testing at less than 20 feet (6 meters).
Pediatric functional muscle testing | 4 weeks
  PFMT will be a useful tool for measurement of muscle strength for children with developmental delay if it be some modifications.
snellen chart for refractive errors | 4 weeks
  The most popular method for assessing visual acuity in clinical settings is still the Snellen chart. A handy tool for rapidly evaluating both monocular and binocular visual acuity is the Snellen chart.

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Iqbal, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schreiber J. Increased intensity of physical therapy for a child with gross motor developmental delay: a case report. Phys Occup Ther Pediatr. 2004;24(4):63-78. doi: 10.1300/j006v24n04_05. PMID 15669670